CLINICAL TRIAL: NCT03708549
Title: Comparison of the Efficacy and Safety of Berberine and Metformin for Schizophrenia Patients With Metabolic Syndrome
Brief Title: Comparison of Berberine and Metformin for the Treatment for MS in Schizophrenia Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ber-Met-MS
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia; Metabolic Syndrome; Berberine; Metformin
Keywords: Berberine; Metformin; Metabolic syndrome; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome | interventions — Berberine; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine group (Experimental): Berberine 300mg（three times a day） plus Metformin simulant 250mg（three times a day）agent plus any atypical antipsychotic drug
  Metformin simulant were matched to metformin in shape, smell and colour were sealed in identical bottles
  Interventions: Drug: Berberine
- Metformin group (Active Comparator): Metformin 250mg（three times a day） plus Berberine simulant 250mg（three times a day）agent plus any atypical antipsychotic drug
  Berberine simulant were matched to Berberine in shape, smell and colour were sealed in identical bottles
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Berberine — The patients will randomly assigned to receive berberine (900 mg day-1, three times a day) and metformin simulant（750mg day-1, three times a day） on the basis of the second-generation antipsychotics monotherapy
  Arms: Berberine group
Drug: Metformin — The patients will randomly assigned to receive metformin (750 mg day-1, three times a day) and berberine simulant（900mg day-1, three times a day） on the basis of the second-generation antipsychotics monotherapy
  Arms: Metformin group

SUMMARY:
Berberine is an isoquinoline alkaloid extracted from medicinal herbs, has been demonstrated to produce beneficial effects on diabetes and hyperlipidemia, fewer study reported its modification on lipid metabolism in schizophrenia. Metformin, have been used for metabolic abnormalities in schizophrenia, findings from these studies indicated that they did have some effect,which are still in experimental stage.This study is aim to compare the efficacy and safety of berberine and metformin for preventing metabolic dysfunction in schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) In accordance with criteria set out in the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV )Axis I Disorders, Clinical Version;
* 2)Meet metabolic syndrome based on Guidelines for Prevention and Treatment of Blood Lipid Abnormality in Chinese Adults(2007);
* 3)Have taken stable dose of the current single antipsychotic drug for at least one month;
* 4) Female subjects will be enrolled to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods during the study.

Exclusion Criteria:

* 1)Individuals who refuse to provide informed consent;
* 2)Currently substance abuse or psychiatrically unstable per treating clinician's judgment;
* 3)One with significant medical illnesses including uncontrolled hypertension, diabetes, seizure disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases also not suitable for this trial;
* 4)Currently on anti-inflammatory or immunosuppressant medication including oral steroids and history of chronic infection (including tuberculosis, HIV and hepatitis), malignancy, organ transplantation, blood dyscrasia, central nervous system demyelinating disorder, and any other known autoimmune or inflammatory condition pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Fasting blood samples for Fasting blood glucose(FBG) | 0, 4, 8,12 weeks
  The main objective is to compare Berberine with Metformin on the effect of reducing the levels of FBG in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of Triglyceride(TG) | 0, 4, 8,12 weeks
  The main objective is to compare Berberine with Metformin on the effect of reducing the levels of TG in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of High-Density Lipoprotein (HDL) | 0, 4, 8,12 weeks
  The main objective is to compare Berberine with Metformin on the effect of reducing the levels of HDL in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of Waist circumference(WC) | 0, 4, 8,12 weeks
  The main objective is to compare Berberine with Metformin on the effect of reducing the levels of WC in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of Blood pressure (BP)，including systolic and diastolic pressure | 0, 4, 8,12 weeks
  The main objective is to compare Berberine with Metformin on the effect of reducing the levels of systolic or diastolic pressure in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment

SECONDARY OUTCOMES:
Changes of Body mass index(BMI) | 0, 4, 8,12 weeks
  Compare Berberine with Metformin on the effect of reducing the levels of BP in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of Positive and Negative Syndrome Scale（PANSS）scores | 0, 4, 8,12 weeks
  Positive and Negative Syndrome Scale（PANSS）has been used to assess symptom severity in schizophrenia.Of the items included in PANSS ,seven constitute a Positive scale,seven form a Negative scale and sixteen constitute a General Psychopathology scale.7-point rating instrument was conceived.A total Score is computed three subscales.Minimum scores is 30 and maximum scores is 210.The higher score are considered the psychiatric symptoms more serious.Compare Berberine with Metformin on the effect of reducing the levels of the scores of PANSS in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of Total Cholesterol(TC) | 0, 4, 8,12 weeks
  Compare Berberine with Metformin on the effect of reducing the levels of TC in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of C reactive protein | 0, 4, 8,12 weeks
  Compare Berberine with Metformin on the effect of reducing the levels of C reactive protein in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment
Changes of Interleukin-1β,Interleukin-6,tumor necrosis factor(TNF-α) | 0, 4, 8,12 weeks
  Compare Berberine with Metformin on the effect of reducing the levels of Interleukin-1β,Interleukin-6,tumor necrosis factor in schizophrenia patients with metabolic syndrome(MS) after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, Tianjin Municipality, China